CLINICAL TRIAL: NCT02758197
Title: The Effects of an Online Mindfulness-Based Stress Reduction (MBSR) Program on Quality of Life and Immune Function Among Cancer Survivors With Chronic Neuropathic Pain
Brief Title: Online MBSR Program for Cancer Survivors With Chronic Neuropathic Pain
Acronym: COMPASSION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20160164-01H
Record Dates: First submitted 2016-04-28; First posted 2016-05-02 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Cancer; Painful Neuropathy; Chronic Pain; Worries; Pain or Disability
Keywords: Mindfulness; Chronic Pain; Quality of Life; Immune Function; Cancer survivors; Disability
MeSH Terms: conditions — Neoplasms; Neuropathy, Painful; Chronic Pain; Pain | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interdisciplinary program including MBSR (Experimental): Participants assigned to this group will be enrolled in an Mindfulness-Based Stress Reduction (MBSR) program following medical treatment optimization. The MBSR program will be composed of eight weekly 2.5 hour sessions and one 6 hour session midway through the course.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)
- Wait-listed Control Group (No Intervention): Participants assigned to this group after medical treatment optimization will act as wait-list controls for the MBSR group. They will be enrolled in the MBSR workshop 3 months after the corresponding intervention group completes the program.

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — Participants assigned to this group will be enrolled in an Mindfulness-Based Stress Reduction (MBSR) course directly following medical treatment optimization. The MBSR course consists of eight weekly 2-hour sessions and one 6 hour session midway through the course and involves psychoeducation, relaxation techniques, gentle stretching (very mild form of yoga), and different forms of meditation. Participants will learn ways to better cope with their pain and the disability and distress related to it with a goal of reducing the stress response that is our body's normal reaction to pain. All sessions will be conducted by a psychologist or social worker with a minimum of 2 years of experience in chronic pain management, formal MBSR training and 2 years of experience leading MBSR groups.
  Other Names: MBSR
  Arms: Interdisciplinary program including MBSR

SUMMARY:
This randomized controlled trial will evaluate the effectiveness of an interdisciplinary treatment approach combining medical management with an online Mindfulness-Based Stress Reduction (MBSR) program in reducing disability and improving quality of life among cancer survivors living with moderate to severe chronic neuropathic pain.

DETAILED DESCRIPTION:
Chronic neuropathic pain (CNP) affects close to 50% of cancer survivors. Even with the best medical treatment, some survivors continue to experience disabling pain. In our recent survey with cancer survivors, we found that the capacity to be aware of different aspects of one's day-to-day experiences, without judgment or reactivity (i.e., being mindful) predicted decreased pain intensity, pain related disability, and increased health-related quality of life among cancer survivors with CNP. Building on these findings, the present randomized controlled trial will evaluate the effectiveness of an online Mindfulness-Based Stress Reduction (MBSR) program for cancer survivors with moderate to severe CNP. The program will benefit patients in rural and remote regions and patients with mobility issues.

We will recruit 100 cancer survivors. All will have their medical treatment optimized by a pain specialist. Additionally, they will complete an 8-week online MBSR program. We hypothesize that the online MBSR program will result in less pain perception, better function and increased health-related quality of life. We will also examine the effects of the MBSR training on biomarkers of stress and immune function.

ELIGIBILITY:
Inclusion Criteria:

* cancer survivors
* experiencing cancer-related neuropathic pain symptoms for at least 3 months
* pain severity ≥4/10 (moderate to severe)
* ability to attend 7 out of 9 MBSR sessions
* ability to complete questionnaires and attend sessions conducted in English or French
* access to the internet and use of an electronic device capable of joining a video conference (i.e., computer or mobile device with a camera and microphone)

Exclusion Criteria:

* expected survival of less than 12 months
* cognitive impairment
* severe psychiatric disorder impacting ability to participate (e.g., schizophrenia, severe depression)
* prior experience with MBSR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-07; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain-related disability, as measured by the Brief Pain Inventory - Pain Interference scale, at 3-month post-intervention. | Baseline and 3 months post-intervention
  The primary outcome is pain-related disability, as measured by the Brief Pain Inventory - Pain Interference scale. The Brief Pain Inventory (BPI) - Pain Interference consists of 7 numerical scales (0 to 10) rating pain interference with general activity, mood, walking ability, work, relations with other people, sleep and enjoyment of life.

SECONDARY OUTCOMES:
Change from baseline in pain severity, as measured by the Brief Pain Inventory - Pain Severity scale, at 3 months post-intervention | Baseline and 3 months post-intervention
  Pain Severity will be measured using the Brief Pain Inventory (BPI) - Pain Severity. The BPI consists of 4 numerical scales (0 to 10) rating pain severity at its worst, at its least, on average, and at the time of filling out the measure. Each severity question is analyzed individually.
Change from baseline in mood states, as measured by the Profile of Mood States scale, at 3 months post-intervention | Baseline and 3 months post-intervention
  The Profile of Mood States (POMS-2A) will be used to measure mood disturbance. Participants are asked to rate 65 adjectives using a 5-point likert scale ( 0= not at all, to 4 = extremely) based on how they have been feeling during the past week, including the day they are filling out the questionnaire. A total mood disturbance score is calculated, as well as scores for 6 sub-scales: depression, tension-anxiety, anger-hostility, vigor-activity, fatigue, confusion-bewilderment.
Overall change in status from baseline, as measured by Patient Global Impression of Change scale, at 3 months post-intervention | Baseline and 3 months post-intervention
  The participants' perceived degree of change in overall status will be measured using the Patient Global Impression of Change (PGIC) scale. The PGIC uses a 7-point likert scale (very much worse, to very much better) to measure how much the participant feels their overall status has changed since the start of the study.
Change from baseline in depressive symptoms, as measured by the Patient Health Questionnaire - 9 scale, at 3 months post-intervention | Baseline and 3 months post-intervention
  The Patient Health Questionnaire - 9 (PHQ-9) is a 9-item scale used to assess the severity of depressive symptoms over the past two weeks and is based on Diagnostic and Statistical Manual (DSM-IV) diagnostic criteria for major depression. Total scores range from 0 to 27, and clinical cut-points correspond to mild, moderate, moderately severe, and severe depression.
Change from baseline in pain catastrophizing, as measured by the Pain Catastrophizing Scale, at 3 months post-intervention. | Baseline and 3 months post-intervention
  The Pain Catastrophizing Scale (PCS) is a 13-item instrument which will evaluate the degree to which patients have negative self-statements and catastrophizing thoughts and ideations when in pain. The PCS uses a 5-point likert scale (0=not at all, 4=all the time) and consists of three subscales (rumination, magnification, helplessness).
Change from baseline in mindfulness, as measured by the Five Facet Mindfulness Questionnaire, at 3 months post-intervention. | Baseline and 3 months post-intervention
  Mindfulness will be measured using the Five Facet Mindfulness Questionnaire (FFMQ). The FFMQ is a 39-item instrument measuring five aspects of mindfulness: Non-reactivity to inner experience, observing, describing, acting with awareness, and non-judging of experience. Participants are asked to use a 5-point Likert-type scale (1 = never or rarely true; 5 = very often or always true) to rate how true of them they believe each statement to be.
Change from baseline in quality of life, as measured by the Functional Assessment of Cancer Therapy - General, at 3 months post-intervention. | Baseline and 3 months post-intervention
  Quality of life will be measured using the Functional Assessment of Cancer Therapy - General (FACT-G). The FACT-G is a 27-item instrument containing general statements which fall within four domains of quality of life: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. Participants are asked to respond to each statement using a 5-point Likert scale from 0 (not at all) to 4 (very much) to indicate how true the statement is for them over the previous seven days.
Change from baseline in fatigue, as measured by the Brief Fatigue Inventory, at 3 months post-intervention. | Baseline and 3 months post-intervention
  Fatigue will be measured using the Brief Fatigue Inventory (BFI). The BFI is a 9-item instrument that measures fatigue severity and the impact it has had on participants' day-to-day functioning in the previous 24 hours. Participants are asked to rate their fatigue at the time of completion as well as their average fatigue and worst fatigue over the previous 24 hours on an 11-point Likert scale from 0 (no fatigue) to 10 (as bad as you can imagine), and the degree to which their fatigue has interfered with their general activity, mood, walking ability, normal work, relations with others, and enjoyment of life over the previous 24 hours on an 11-point Likert scale from 0 (does not interfere) to 10 (completely interferes).
Change from baseline in fear of cancer recurrence, as measured by the Fear of Cancer Recurrence Inventory, at 3 months post-intervention. | Baseline and 3 months post-intervention
  Fear of cancer recurrence will be measured using the Fear of Cancer Recurrence Inventory (FCRI). The FCRI is a 42-item instrument that measures seven factors of cancer recurrence: triggers, severity, psychological distress, functional impairment, insight, reassurance, and coping strategies. Participants respond to questions using a 5-point Likert scale from 0 (not at all or never) to 4 (a great deal or all the time). The scale provides a global score as well as seven sub-scale scores; one for each factor. A higher score indicates higher levels of fear of cancer recurrence.
Change from baseline in immune function, as measured by blood levels of tumor necrosis factor - alpha interleukin-6, interleukin-4, interleukin-10, and c-reactive protein at 3 months post-intervention. | Baseline and 3 months post-intervention
  Immune function, with particular attention to the following parameters: tumor necrosis factor - alpha (TNF-α), interleukin-6 (IL-6), interleukin-4 (IL-4), interleukin-10 (IL-10), and c-reactive protein (CRP) will be measured from participant blood samples. Six mL whole blood samples will be obtained from participants and the concentration of these parameters will be quantified and recorded. All samples and standards will be analyzed in duplicate.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Poulin, Ph.D, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No